CLINICAL TRIAL: NCT04851366
Title: Selective PRevention Through transdiagnOstiC Intervention for Adolescents at Risk of Emotional Disorders (PROCARE)
Brief Title: Selective Prevention Transdiagnostic Intervention for At-risk Adolescents
Acronym: PROCARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Collaborators: Universidad Miguel Hernandez de Elche (Other); University Rovira i Virgili (Other); University of Miami (Other)
Responsible Party: Principal Investigator, LuisJoaquin Garcia-Lopez, Professor, University of Jaén
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: PID2019-111138RB-I00
Record Dates: First submitted 2021-04-11; First posted 2021-04-20 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Anxiety Disorders and Symptoms; Depressive Symptoms
Keywords: ADOLESCENCE; TRANSDIAGNOSTIC; SELECTIVE PREVENTION; Randomized-Controlled Trial; AT-RISK
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Two interventions are evaluated in parallel against a active control group
Who Masked: Participant, Outcomes Assessor
Masking Description: A three-armed simple-blind RCT will be conducted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PROCARE+ (with add-on modules) (Experimental): In addition to core UP-A preventive intervention, PROCARE will apply an innovative personalized medicine approach by adding specific modules according to the risk factor evidenced by adolescents. Different modules will be suited for the stratified groups in a more personalized format. Add-on young-focused modules would include, but not limited to social, parental, stress-related (including CoVid19 impact) risk factors, and health. Dosage (number of modules) will be included as covariate in all subsequent analyses.
  Interventions: Behavioral: PROCARE+ (with add-on modules)
- PROCARE (UP-A for selective purposes) (Experimental): To ensure cost-effectiveness, PROCARE core intervention will be designed as a brief 8-session child-focused programme which aims to build resilience for adolescents by adapting the core modules from UP-A, along with one individual session with adolescent and parents. Sessions will be delivered in reduced groups, using a typical selective preventive intervention format focused on cost-effectiveness.
  Interventions: Behavioral: PROCARE (UP-A for selective purposes)
- Active control condition. (Active Comparator): The active control condition will be based on the "U talk programme" developed by Prf. Jill Ehrenreich-May at University of Miami and colleagues. It follows a similar structure as the UP-A original programme and allows for two alternative compare conditions to PROCARE. The U Talk programme support-based group condition will be used as active control condition.
  Interventions: Behavioral: Active control condition

INTERVENTIONS:
Behavioral: PROCARE+ (with add-on modules) — The modules will mainly consist in therapy sessions to provide the adolescents with tools to confront risk situations such as communication skills, coping skills to manage stress, etc. The group will include education about discussing thoughts, feelings, and behaviour as parts of emotion, and emphasis on providing support around the specific risks factors detected.
  Arms: PROCARE+ (with add-on modules)
Behavioral: PROCARE (UP-A for selective purposes) — This core intervention is meant to respond to the heterogeneity inherent in emotional difficulties presentation by extinguishing distress associated with the presentation of heightened negative emotion in general and reduction or elimination of resultant emotionally-driven behaviours, including avoidance, escape, aggression, and controlling behaviours (e.g., reassurance seeking) that reinforce emotional distress intensity over time.
  Arms: PROCARE (UP-A for selective purposes)
Behavioral: Active control condition — Psychoeducation about many different emotions, emphasis on discussing thoughts, feelings, and behavior as parts of emotion, and emphasis on providing support around generally distressing events.
  Arms: Active control condition.

SUMMARY:
Emotional disorders (anxiety and/or depression) are severely undiagnosed and untreated despite being among the most common mental disorders, particularly at a young age. Half of all mental disorders begin by age 14; three-quarters by age 24, which makes adolescence a particularly crucial stage. In adolescence, prodromal signs of mental disorders and even full-blown clinical conditions often remain undetected, undiagnosed and untreated. However, there is an absence of evidence-based protocols to reach at-risk youth for developing emotional disorders. There is an urgent need for a paradigm shift by developing intervention protocols to early identify and treat at-risk adolescents, thus preventing them from developing severe mental disorders later on in life. Mental health selective prevention is key to helping at-risk adolescents thrive before emotional disorder evolves. To cover this gap, PROCARE is conceptualized as a modularized selective preventive programme for adolescents aged 12 to 18 years. Using personalized medicine approach, PROCARE will allow to tailor intervention protocols according to the particular needs of an individual, but also to identify vulnerable people according to risk factors. Adolescents will be stratified based on risk and resilience status and allocated to a 3-arm intervention trial, delivered as a group, face-to-face or telehealth format, depending on Covid19 restrictions imposed by government. By the very first time, PROCARE as selective intervention for at-risk adolescents will deliver specific add-on modules to tackle risk factors evidenced by adolescents, along with a core intervention. The PROCARE protocol aims to reduce the effect of risk factors and enhance protective factors that will eventually lead to lasting positive effects for adolescents. PROCARE will combine quantitative analysis, with special attention to vulnerable groups in a sex/gender disaggregated way. The PROCARE project is expected to have a far impact ultimately contributing to preventing and reducing the prevalence of mental disorders in the young. The outcomes of PROCARE will contribute to identifying and treating adolescents at risk for emotional mental at an early stage, before they incur personal, societal and economic cost. PROCARE will be culturally-adapted and implemented as a multicenter Randomized-Controlled Trial (RCT). PROCARE will be designed to be an acceptable, scalable, and sustainable selective prevention program.

DETAILED DESCRIPTION:
OBJECTIVES The general objective of PROCARE is to design, implement and evaluate a selective preventive intervention for adolescents aged 12-18 at risk of emotional disorders like anxiety and depression. The core intervention will be based on the Unified protocol for transdiagnostic treatment of emotional disorders in adolescents (UP-A), already proven as effective in the US, but adapted with selective prevention purposes thanks support of main author of the protocol (Prf. Ehrenreich-May). By the very first time, PROCARE as selective intervention for at-risk adolescents will deliver specific add-on modules to tackle risk factors evidenced by adolescents. So, PROCARE will be flanked with a preliminary risk and resilience factor stratification, according to the identified users' and stakeholders' needs in order to empower emotional regulation, building resilience and coping capacities. It will be culturally-adapted and designed to be an acceptable, scalable, and sustainable selective prevention program.

The specific objectives of the PROCARE project are:

* To identify adolescents at risk for emotional difficulties via a thorough screening risk and resilience factor analysis. The personalised medicine approach will allow the team to tailor add-on intervention modules according to the particular needs of every subject but also to know what risk factors are the best indicators to identify young people at risk and/or indicators of the effectiveness of the programme.
* To implement a selective preventive transdiagnostic intervention for adolescents at risk of developing mental health problems like anxiety and depression that will serve as a gold standard in the field. The preventive programme will be adapted from the UP-A protocol for clinical population; tailoring it to the specific requirements of recruited adolescents with add-on modules according to the risk factors presented. Thanks to the support of a strong External Advisory Board (EAB): Asociación Española de Ayuda Mutua contra Fobia Social y Trastornos de Ansiedad (AMTAES), Federación Estatal de Lesbianas, Gais, Trans y Bisexuales (FELGTB), Instituto de la Juventud (INJUVE/Spanish MInistry of Social Affairs and Agenda 2030) & Confederación de Organizaciones de Psicopedagogía y Orientación de España (COPOE), PROCARE will be designed to be an acceptable, scalable, and sustainable face-to-face selective prevention program for use in culturally-diverse school setting, avoiding stigmatization or via telehealth, depending on governmental restrictions due to pandemia.
* To demonstrate cost-effectiveness of the intervention using a rigorous scientific method. Designed as a three-arm RCT (Arm 1 = Active Control group; Arm 2 = PROCARE without add-on modules (UP-A adapted for selective prevention); Arm 3 = PROCARE with add-on modules;) and a baseline, post-test, 6-month and one-year follow-up, PROCARE will meet internationally adopted guidelines to maximise the reliability of results in preventive trials.
* To facilitate the replication of the programme based on a well-defined methodology and analysis plan and elaborate practice guidelines for mental health problems amongst adolescents. These guidelines will be used as a gold standard for prevention. The evaluation will combine quantitative and qualitative methods and the analysis of the findings: (a) in a qualitative way, (b) in a quantitative way and (c) in a sex disaggregated way, by examining differences between boys and girls and data intersecting with sex (cultural gender norms and emotion regulation skills) that can help to explain these differences.

The preventive approach outlined in PROCARE is aimed at serving as a blueprint to timely detect and intervene in young people at risk and to contribute to the promotion of emotional mental health in the young.

The PROCARE project will bundle the resources for the improvement of health and wellbeing at early ages. This action will be focused on preventing emotional problems by a sequenced approach to skill development, resilience, an explicit implementation guidelines and effective training to mental health providers.

METHODOLOGY The methodology was designed in order to achieve the project's objective of presenting a novel approach to treating adolescents at risk of developing emotional disorders, in response to current trends for selective prevention and personalized medicine. PROCARE working plan will be divided into 3 interconnected stages. Firstly, in order to identify adolescents at risk of suffering emotional disorders (anxiety and depression), the following self-reports will be administered to adolescents: Strengths and Difficulties Questionnaire (SDQ) to evaluate adolescents at-risk of emotional disorders, the Connor-Davidson Resilience Scale (CD-RISC) to assess resilience, and the Revised Child Anxiety and Depression Scale-30 (RCADS-30) will screen for presence/absence of emotional symptomatology. Second, putative risk factors will be collected by adolescents, parents and teachers in those adolescents who are retained. These factors will serve for stratification for tailoring add-on intervention modules according to the particular needs of every subject but also to know which risk factors are the best indicators to: (i) identify subjects at risk, (ii) predict response to the selective preventive intervention (PROCARE) and to (iii) define short- and long-term mechanisms of action of the selective preventive intervention (PROCARE). Valuing voices from stakeholders and end-users, the investigators will focus on the study of the influence of the above-described variables. Third, the investigators will test a selective preventive intervention using multi-center randomized control trial and personalised medicine approach. Special attention will be paid to particularly vulnerable young people, such as disabled, refugees, immigrants, or minorities (national, ethnic, linguistic, religious, and sexual).

IMPACT The need to include mental health among the first priorities of the public health agenda has been increasingly recognized over the past decades. The outcomes of the PROCARE project will have a far impact ultimately contributing to preventing and reducing the prevalence of mental disorders in the young. These problems are wide-ranging, long-lasting, and enormous and impose a range of costs on individuals, families and communities. The outcomes of the project, if successful, will have far reaching implications, contributing to identifying and treating adolescents at risk for emotional mental at an early stage, before they incur personal, societal and economic cost.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent from adolescent and legal guardian
* able to attend prevention modules on his/her own
* Strengths and Difficulties Questionnaire "unlikely" or "possible diagnoses"
* score on Connor-Davidson Resilience Scale as low or medium resilient,
* score below cut-off for Revised Child Anxiety and Depression Scale-30
* evidence of risk factors (social exclusion, stress-related situations, unhealthy lifestyle habits, parental-child interaction)
* absence of anxiety and/or mood disorders
* not receiving psychological or psychiatric treatment
* not presenting acute suicidality and (9) absence of neurodevelopmental disorders.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 208 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Factors associated with adolescents' mental health | Baseline to 12 months after start of interventions
  The study's primary outcome was self-reported risk and protective factors level of emotional disorders as assessed by Strengths and Difficulties Questionnaire (SDQ). Total scores range from 0 to 50. Higher scores mean a worse outcome.
Resilience | Baseline to 12 months after start of interventions
  Self-reported resilience, as measured by Connor-Davidson Resilience Scale (CD-RISC). Total scores range from 0 to 100. Higher scores mean a better outcome.
Health-related quality of life | Baseline to 12 months after start of interventions
  Secondary outcome assessed included self-reported changes in health-related quality of life as assessed by KIDSCREEN-10. Total scores range from 10 to 50. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Emotion regulation skills | Baseline to 12 months after start of interventions
  Emotion regulation skills as assessed by Difficulties in Emotion Regulation Scale-36 (DERS-36). Total scores range from 36 to 180. Higher scores mean a worse outcome.
Psychological flexibility | Baseline to 12 months after start of interventions
  Psychological flexibility as assessed by Willingness and Action Measure for Children and Adolescents (WAM-C/A). Total scores range from 0 to 56. Higher scores mean a better outcome.
Self-reported anxiety and mood symptomatology | Baseline to 12 months after start of interventions
  The study's primary outcome was self-reported anxiety and mood symptomatology as assessed by Revised Child Anxiety Depression Scale (RCADS-30). Total scores range from 0 to 90. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: LuisJoaquin Garcia-Lopez, PhD, Principal Investigator — University of Jaen
Locations (3):
- Spain (3):
  - Universidad Miguel Hernandez, Elche, Alicante
  - University of Jaen, Jaén, Jaen
  - Universitat Rovira i Virgili, Tarragona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Garcia-Escalera J, Valiente RM, Sandin B, Ehrenreich-May J, Prieto A, Chorot P. The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Adolescents (UP-A) Adapted as a School-Based Anxiety and Depression Prevention Program: An Initial Cluster Randomized Wait-List-Controlled Trial. Behav Ther. 2020 May;51(3):461-473. doi: 10.1016/j.beth.2019.08.003. Epub 2019 Aug 14. PMID 32402261
- [Result] Sandin B, Garcia-Escalera J, Valiente RM, Espinosa V, Chorot P. Clinical Utility of an Internet-Delivered Version of the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Adolescents (iUP-A): A Pilot Open Trial. Int J Environ Res Public Health. 2020 Nov 10;17(22):8306. doi: 10.3390/ijerph17228306. PMID 33182711
- [Result] Levin L, Henderson HA, Ehrenreich-May J. Interpersonal predictors of early therapeutic alliance in a transdiagnostic cognitive-behavioral treatment for adolescents with anxiety and depression. Psychotherapy (Chic). 2012 Jun;49(2):218-230. doi: 10.1037/a0028265. PMID 22642525
- [Result] Queen AH, Barlow DH, Ehrenreich-May J. The trajectories of adolescent anxiety and depressive symptoms over the course of a transdiagnostic treatment. J Anxiety Disord. 2014 Aug;28(6):511-21. doi: 10.1016/j.janxdis.2014.05.007. Epub 2014 Jun 2. PMID 24960439
- [Result] Bilek EL, Ehrenreich-May J. An open trial investigation of a transdiagnostic group treatment for children with anxiety and depressive symptoms. Behav Ther. 2012 Dec;43(4):887-97. doi: 10.1016/j.beth.2012.04.007. Epub 2012 May 1. PMID 23046789
- [Result] Ehrenreich-May J, Rosenfield D, Queen AH, Kennedy SM, Remmes CS, Barlow DH. An initial waitlist-controlled trial of the unified protocol for the treatment of emotional disorders in adolescents. J Anxiety Disord. 2017 Mar;46:46-55. doi: 10.1016/j.janxdis.2016.10.006. Epub 2016 Oct 17. PMID 27771133